CLINICAL TRIAL: NCT07273006
Title: Percutaneous Electrical Nerve Stimulation As Alternative To Nerve Blocks In Anesthesia, Pain Medicine And Rehabilitation Of Nonspecific Chronic Pain
Acronym: PENSAR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Universidad Francisco de Vitoria (Other); Medical University of Warsaw (Other); Jagiellonian University (Other)
Responsible Party: Principal Investigator, JUAN ANTONIO VALERA CALERO, Doctor in Health Sciences, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UComplutenseMadrid-PENSAR
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non-specific Low Back Pain (NSLBP); Facet Joint Syndrome
Keywords: musculoskeletal ultrasound imaging; health care cost-utility; safety and adverse events; randomized clinical trial; pain neuromodulation; diagnostic nerve blocks; percutaneous electrical nerve stimulation; facet joint syndrome; non-specific low back pain
MeSH Terms: interventions — Nerve Block; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor would be a different investigator blinded to the interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PENS (Experimental): A single ultrasound-guided session will be applied using fine solid needles (0.32 mm diameter), accounting for dual innervation. Electrical parameters will be fixed within recommended ranges (10 Hz, 250 µs, current intensity sufficient to produce a strong but tolerable sensation below the motor threshold using a standardized ramp, and session duration of 20 minutes).
  Interventions: Device: Percutaneous electrical nerve stimulation
- Nerve block (Active Comparator): Two adjacent levels per joint will be blocked in a single session. After minimal intradermal infiltration for local anesthesia, a sterile 25G-22G needle will be inserted in-plane toward the target under continuous visualization. Before administering the drug in opaque syringes, negative aspiration and fractional injection will be performed, confirming the absence of abnormal resistance or radiating pain. The diagnostic injectate will be a local anesthetic without corticosteroid (1% lidocaine) with low volumes of 0.5 ml per branch to limit diffusion.
  Interventions: Drug: Nerve block with Lidocain
- PENS + nerve block (Active Comparator): Both procedures will be performed in a single visit (first PENS, followed by the nerve block) following the same procedures described above
  Interventions: Drug: Nerve block with Lidocain; Device: Percutaneous electrical nerve stimulation
- PENS + placebo block (Sham Comparator): In the same visit, PENS will be applied following the same described protocol, and the full ritual of the nerve block will be reproduced. However, in this group, no active drug will be administered (a minimal volume of inert solution will be injected into the subcutaneous/superperiosteal plane to mimic the injection sensation without depositing perineural anesthetic).
  Interventions: Device: Percutaneous electrical nerve stimulation; Other: Sham Block

INTERVENTIONS:
Drug: Nerve block with Lidocain — Two adjacent levels per joint will be blocked in a single session. After minimal intradermal infiltration for local anesthesia, a sterile 25G-22G needle will be inserted in-plane toward the target under continuous visualization. Before administering the drug in opaque syringes, negative aspiration and fractional injection will be performed, confirming the absence of abnormal resistance or radiating pain. The diagnostic injectate will be a local anesthetic without corticosteroid (1% lidocaine) with low volumes of 0.5 ml per branch to limit diffusion
  Arms: Nerve block; PENS + nerve block
Device: Percutaneous electrical nerve stimulation — A single ultrasound-guided session will be applied using fine solid needles (0.32 mm diameter), accounting for dual innervation. Electrical parameters will be fixed within recommended ranges (10 Hz, 250 µs, current intensity sufficient to produce a strong but tolerable sensation below the motor threshold using a standardized ramp, and session duration of 15-20 minutes)
  Arms: PENS; PENS + nerve block; PENS + placebo block
Other: Sham Block — The full ritual of the nerve block will be reproduced. However, in this group, no active drug will be administered (a minimal volume of inert solution will be injected into the subcutaneous/superperiosteal plane to mimic the injection sensation without depositing perineural anesthetic)
  Arms: PENS + placebo block

SUMMARY:
Chronic musculoskeletal pain of non-specific origin affects approximately 30% of the global population. Beyond its prevalence, it represents a serious health and socioeconomic problem. It is considered the leading cause of years lived with disability and is characterized by persistent functional limitation, deterioration of quality of life, and poorer mental health, with a high comorbidity of depression, anxiety, and sleep disorders, as well as a greater risk of suicidal ideation and behavior.

From a socioeconomic perspective, chronic pain entails an impact of up to USD 635 billion annually just in United States (USA). In fact, spinal pain alone represents the condition with the highest direct costs (around USD 134.5 billion in USA) and additional indirect costs due to absenteeism and presenteeism, which impair productivity and work performance. These figures are expected to be substantially higher when considered at a global scale.

One of the main aggravating factors of this condition is that in up to 90% of patients experiencing pain there is no identifiable anatomopathological substrate that reliably explains the symptoms (non-specific pain). Radiological findings are extremely common in asymptomatic populations, and making diagnostic or therapeutic decisions based on such findings, promotes overdiagnosis and low-value clinical cascades. It is estimated that up to 50% of imaging requests and 60% of spinal surgeries6 are unnecessary or unjustified. For this reason, Clinical Practice Guidelines recommend prioritizing interventional diagnostic techniques based on functional criteria over the interpretation of radiological findings, as they allow for more sensitive and specific identification of nociceptive sources (with a recommendation grade I-II).

In this context, the motivation of the project is to study PENS as a non-pharmacological, safe, and transferable alternative to nerve blocks, reducing the risk of complications associated with the use of local anesthetics/corticosteroids and large-gauge needles. According to recent systematic reviews and meta-analyses confirming immediate analgesic responses, PENS could be a feasible alternative that maintains functional diagnostic and therapeutic value with a generally mild adverse-event profile and lower cost.

DETAILED DESCRIPTION:
Within the broad spectrum of chronic pain conditions, low back pain (LBP) is the leading cause of years lived with disability worldwide and one of the largest contributors to the global disease burden. According to the latest Global Burden of Disease analysis, approximately 620 million people suffered from LBP in 2020. Projections for the coming decades are not encouraging since, by 2050, the number of affected individuals is expected to rise to 843 million, a 36.4% increase compared to 2020. This growth will be mainly driven by population increase and aging, with the sharpest rises expected in Asia and Africa.

Beyond its direct health consequences, LBP imposes a considerable economic burden on both individuals and societies, as its highest incidence occurs during the most productive working years (approximately 45-55 years old). In the USA alone, direct costs related to spinal disorders reached USD 315 billion between 2012 and 2014, in addition to productivity losses estimated in hundreds of millions of workdays each year. Considering its growing prevalence and socioeconomic implications, LBP is regarded as a global health priority.

LBP may originate from a wide variety of musculoskeletal, neurological, or visceral conditions, and its clinical expression may combine nociceptive mechanisms (related to tissue injury or stimulation of lumbar structures), neuropathic mechanisms (involving lesions or disease of the somatosensory system), and nociplastic mechanisms (involving altered nociceptive processing without structural lesions, often with central sensitization and descending inhibitory dysfunction).

Current clinical frameworks establish that in up to 90% of patients, it is not possible to identify a clear anatomopathological pain source (thus defined as non-specific LBP). The main challenge lies in identifying which structures (i.e., intervertebral discs, facet /zygapophyseal joints, sacroiliac joints, ligaments, or myofascial tissues) are the nociceptive sources. The absence of a defined structural correlate (as most structural abnormalities are also frequent in asymptomatic individuals) largely explains the high recurrence and chronicity rates, as well as the frequency of ineffective treatments, unjustified surgeries, and the economic impact of healthcare utilization without a clearly established etiology. Consequently, diagnosis in these patients is essentially clinical and based on exclusion criteria, with a therapeutic focus on symptom modulation and functional recovery rather than on identifying and correcting a single structural lesion.

Although scientific evidence consistently supports the high percentage of non-specific LBP cases and discourage routine imaging in such patients, this practice remains common in hospital care. It is estimated that 30% to 55% of imaging studies requested for LBP are unnecessary or not clinically indicated. The indiscriminate use of imaging not only generates unnecessary costs and delays, but also exposes patients to unjustified radiation and overdiagnosis risk. For example, the prevalence of disc protrusions in asymptomatic individuals increases from 30% at age 20 to 84% at age 80, which may lead to misinterpreting benign degenerative changes as pathological, fueling overtreatment and patient anxiety.

Consequently, this practice directly impacts the high rate of unnecessary spinal surgeries. It is estimated that up to 60% of spinal surgeries are performed unnecessarily, without clear indications, neurological deficits, or relevant radiographic findings. These procedures not only expose patients to avoidable risks with limited effectiveness, but also represent an annual cost of USD 4 billion in the USA.

In the absence of clinical or radiological criteria with sufficient diagnostic precision, international clinical practice guidelines, such as those of the American Society of Interventional Pain Physicians, recommend diagnostic anesthetic blocks as the reference procedure to confirm the nociceptive source (with evidence level I-II and moderate to strong recommendation strength). These diagnostic blocks consist of controlled injections of local anesthetics to determine the involvement of specific structures depending on the patient's pain relief response. For example, the facet joint can be functionally identified as the pain source through controlled infiltration of local anesthetic into the medial branches of the dorsal rami that innervate the lumbar facets. If a transient and reproducible analgesic response occurs after the block (particularly when comparative blocks with anesthetics of different duration are used) the diagnosis of facet joint syndrome is confirmed, supporting the appropriateness of subsequent interventions.

Despite their strong recommendation level, these procedures are not free of complications and risks, associated with large-gauge needles and local anesthetic administration. Common complications include peripheral nerve injury from direct mechanical trauma, intrafascicular injection, ischemia, or anesthetic neurotoxicity, with reported incidences of transient neuropathic symptoms ranging from 0% to 41%, and permanent injury below 1%. Other potential complications include systemic toxicity of local anesthetics (potentially severe if intravascular injection occurs), local infection or abscess formation, and, less frequently, nerve compression due to fibrosis or hematoma. Risk factors such as middle age (40-65 years), smoking, pre-existing neuropathy, or metabolic diseases (e.g., diabetes, chronic obstructive pulmonary disease) increase susceptibility to neural damage. Although ultrasound-guided techniques have substantially reduced the risk of major events, they do not eliminate the possibility of post-block neuropathies or adverse anesthetic reactions.

PENS constitutes a minimally invasive alternative that avoids corticosteroids and anesthetics, reduces exposure to large-volume injectables, and produces reproducible analgesic responses, useful as a functional test supporting the diagnostic hypothesis, while also serving as a therapeutic option within a multimodal pain management approach. This technique applies low- or high-frequency electrical currents (2-100 Hz) via fine needles, aiming to activate large-diameter myelinated afferent fibers and modulate nociceptive transmission at the spinal level. It has been shown to induce endogenous analgesic mechanisms through opioid neurotransmitter (µ, δ, κ) release and activation of descending inhibitory pathways, reducing central sensitization and improving conditioned pain modulation. These neurophysiological effects explain its capacity to reduce primary and secondary hyperalgesia observed in chronic musculoskeletal syndromes, particularly in the short term. Indeed, systematic reviews and meta-analyses report that PENS reduces pain and disability compared to placebo and other interventions.

These properties suggest that PENS may represent a feasible and safe alternative to anesthetic blocks for modulating facet-origin lumbar pain, offering an option that eliminates the risks associated with drugs used in blocks (e.g., systemic toxicity of local anesthetics, allergic reactions, systemic corticosteroid effects, hyperglycemia, adrenal suppression) by not requiring substance injection. From a mechanical perspective, PENS uses solid fine-gauge needles (≈0.25-0.30 mm; 32-34G), significantly thinner than those typically used for medial branch blocks (≈22-25G; 0.5-0.7 mm), thereby reducing tissue trauma, hematoma risk, and nerve injury probability. The absence of injectables also decreases the risk of local anesthetic systemic toxicity and prevents intra-articular or perineural pressure increases.

In terms of practical safety, adverse events with PENS are usually mild and self-limited (transient localized pain, small bruising, occasional vasovagal reactions), with a particularly favorable profile in patients with comorbidities where blocks carry higher risk (e.g., poorly controlled diabetes, prior adverse reactions to anesthetics, or contraindications to corticosteroids). With aseptic technique and ultrasound guidance when appropriate, PENS offers a minimally invasive alternative that preserves the diagnostic/therapeutic modulation capability over the facet target, while substantially reducing pharmacological and mechanical risks associated with conventional blocks.

Therefore, the general objective is to evaluate PENS as a diagnostic alternative not inferior to nerve blocks and as a therapeutic modality in chronic LBP of suspected facet origin, to establish its optimal dosage, and to assess its safety, resource utilization, and cost-utility in multicenter outpatient settings.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic LBP lasting at least three months and clinical suspicion of facet joint pain.
* A balanced sex distribution and a wide range of body mass index (BMI) will be promoted to allow subgroup analyses and to explore potential associations between obesity and procedural complications, thus strengthening the external validity of the study. This demographic selection is justified by prevalence patterns reported in the literature and by the need to capture clinically relevant effect modifiers in real clinical environments.
* The suspicion of facet joint pain will be based on a compatible axial clinical pattern and the absence of objective neurological deficit, considering that neither physical examination nor imaging tests provide sufficient specificity. Therefore, diagnostic confirmation will be performed functionally through ultrasound-guided medial branch diagnostic blocks, which are the most reliable tool for attributing pain to the facet joint. The dual innervation of each lumbar facet joint will be considered; thus, two adjacent levels will be blocked per joint (the medial branch at the affected level and the one immediately above).
* Eligible patients will be those with a positive functional screening in two independent medial branch diagnostic blocks performed with anesthetics of different duration, in separate sessions, to reduce false positives.
* The diagnosis will be confirmed in cases reporting clinically relevant pain relief within the expected pharmacological window.

Exclusion Criteria:

* Exclusion criteria will include red flags or specific etiologies such as infection, neoplasm, fracture, or cauda equina syndrome, as well as patients with progressive motor radiculopathy or another demonstrated neuropathic pain source other than facet origin.
* Individuals who have undergone prior procedures that could compromise response interpretation such as recent radiofrequency denervation, cryoneurolysis or intra-articular corticosteroid injections within a period that could extend analgesic effects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | From baseline within the pre-specified time window for each intervention (two post-intervention assessments will be performed in all groups at 15 and 45 minutes) and maintained at 7 days
  The primary variable will be immediate analgesic response, defined as a ≥50% reduction in the Numerical Pain Rating Scale (NPRS, 0-10). Lower scores indicate less pain intensity.

SECONDARY OUTCOMES:
Pain during specific movements | Baseline, 45 minutes, and 7 days
  Participants will be asked to rate, using the Numerical Pain Rating Scale (NPRS) from 0-10 (lower scores indicate less pain intensity), their pain during lumbar flexion, rotation, extension and inclination
Pressure pain threshold | Baseline, 45 minutes, and 7 days
  An algometer will be used to determine the mechanosensitivity over the projection of the symptomatic facet joint.
Analgesic drug consumption | From 3 months before the study until 7 days after the intervention.
  A record will be used.
Participants' satisfaction | After 7 days
  Patients will be asked to rate in a 0-10 scale their satisfaction with the intervention.

OTHER OUTCOMES:
Record of local and systemic adverse events | Baseline, 7 days
  Any adverse events or sequelae (defined as short-medium term symptoms perceived as unacceptable by the patient or that required further treatment) experienced during or 7 days after the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Valera-Calero, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Medical University of Warsaw, Warsaw, Warszawa, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Valera-Calero JA, Plaza-Manzano G, Rabanal-Rodriguez G, Diaz-Arribas MJ, Kobylarz MD, Buffet-Garcia J, Fernandez-de-Las-Penas C, Navarro-Santana MJ. Current State of Dry Needling Practices: A Comprehensive Analysis on Use, Training, and Safety. Medicina (Kaunas). 2024 Nov 14;60(11):1869. doi: 10.3390/medicina60111869. PMID 39597054
- [Result] Rabanal-Rodriguez G, Navarro-Santana MJ, Valera-Calero JA, Gomez-Chiguano GF, Kocot-Kepska M, Fernandez-de-Las-Penas C, Plaza-Manzano G. Neurophysiological Effects of Dry Needling: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2025 Sep 6:S0003-9993(25)00887-1. doi: 10.1016/j.apmr.2025.08.019. Online ahead of print. PMID 40921318
- [Result] Mogedano-Cruz S, Lopez-Perez M, Gijon-Lago D, Romero-Morales C, Alonso-Perez JL, Villafane JH, Saiz SLJ, Sosa-Reina MD. Peripheral Percutaneous Electrical Nerve Stimulation for Neuropathies: A Systematic Review and Meta-analysis. Pain Manag Nurs. 2025 Feb;26(1):93-101. doi: 10.1016/j.pmn.2024.11.005. Epub 2024 Dec 13. PMID 39674759
- [Result] Phan KH, Anderson JG, Bohay DR. Complications Associated with Peripheral Nerve Blocks. Orthop Clin North Am. 2021 Jul;52(3):279-290. doi: 10.1016/j.ocl.2021.03.007. Epub 2021 May 7. PMID 34053573
- [Result] Hall AM, Aubrey-Bassler K, Thorne B, Maher CG. Do not routinely offer imaging for uncomplicated low back pain. BMJ. 2021 Feb 12;372:n291. doi: 10.1136/bmj.n291. No abstract available. PMID 33579691
- [Result] Chou R, Fu R, Carrino JA, Deyo RA. Imaging strategies for low-back pain: systematic review and meta-analysis. Lancet. 2009 Feb 7;373(9662):463-72. doi: 10.1016/S0140-6736(09)60172-0. PMID 19200918
- [Result] GBD 2021 Low Back Pain Collaborators. Global, regional, and national burden of low back pain, 1990-2020, its attributable risk factors, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 May 22;5(6):e316-e329. doi: 10.1016/S2665-9913(23)00098-X. eCollection 2023 Jun. PMID 37273833
- [Result] Plaza-Manzano G, Gomez-Chiguano GF, Cleland JA, Arias-Buria JL, Fernandez-de-Las-Penas C, Navarro-Santana MJ. Effectiveness of percutaneous electrical nerve stimulation for musculoskeletal pain: A systematic review and meta-analysis. Eur J Pain. 2020 Jul;24(6):1023-1044. doi: 10.1002/ejp.1559. Epub 2020 Apr 4. PMID 32171035
- [Result] Olivier TJ, Konda C, Pham T, Baltich Nelson B, Patel A, Sharma GS, Trivedi K, Annaswamy TM. Clinical practice guidelines on interventional management of low back pain: A synthesis of recommendations. PM R. 2023 Aug;15(8):1052-1063. doi: 10.1002/pmrj.12930. PMID 36507598
- [Result] Busse JW, Genevay S, Agarwal A, Standaert CJ, Carneiro K, Friedrich J, Ferreira M, Verbeke H, Brox JI, Xiao H, Virdee JS, Gunderson J, Foster G, Heegsma C, Samer CF, Coen M, Guyatt GH, Wang X, Sadeghirad B, Malam F, Zeraatkar D, Vandvik PO, Zhou T, Xie F, Siemieniuk RAC, Agoritsas T. Commonly used interventional procedures for non-cancer chronic spine pain: a clinical practice guideline. BMJ. 2025 Feb 19;388:e079970. doi: 10.1136/bmj-2024-079970. PMID 39971339
- [Result] Manchikanti L, Kaye AD, Soin A, Albers SL, Beall D, Latchaw R, Sanapati MR, Shah S, Atluri S, Abd-Elsayed A, Abdi S, Aydin S, Bakshi S, Boswell MV, Buenaventura R, Cabaret J, Calodney AK, Candido KD, Christo PJ, Cintron L, Diwan S, Gharibo C, Grider J, Gupta M, Haney B, Harned ME, Helm Ii S, Jameson J, Jha S, Kaye AM, Knezevic NN, Kosanovic R, Manchikanti MV, Navani A, Racz G, Pampati V, Pasupuleti R, Philip C, Rajput K, Sehgal N, Sudarshan G, Vanaparthy R, Wargo BW, Hirsch JA. Comprehensive Evidence-Based Guidelines for Facet Joint Interventions in the Management of Chronic Spinal Pain: American Society of Interventional Pain Physicians (ASIPP) Guidelines Facet Joint Interventions 2020 Guidelines. Pain Physician. 2020 May;23(3S):S1-S127. PMID 32503359
- [Result] AlAli KF. Unnecessary spine surgery: can we solve this ongoing conundrum? Front Surg. 2023 Aug 25;10:1270975. doi: 10.3389/fsurg.2023.1270975. eCollection 2023. No abstract available. PMID 37693642
- [Result] Logan GS, Pike A, Copsey B, Parfrey P, Etchegary H, Hall A. What do we really know about the appropriateness of radiation emitting imaging for low back pain in primary and emergency care? A systematic review and meta-analysis of medical record reviews. PLoS One. 2019 Dec 5;14(12):e0225414. doi: 10.1371/journal.pone.0225414. eCollection 2019. PMID 31805073
- [Result] Jenkins HJ, Downie AS, Maher CG, Moloney NA, Magnussen JS, Hancock MJ. Imaging for low back pain: is clinical use consistent with guidelines? A systematic review and meta-analysis. Spine J. 2018 Dec;18(12):2266-2277. doi: 10.1016/j.spinee.2018.05.004. Epub 2018 May 3. PMID 29730460
- [Result] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Result] de Luca K, Tavares P, Yang H, Hurwitz EL, Green BN, Dale H, Haldeman S. Spinal Pain, Chronic Health Conditions and Health Behaviors: Data from the 2016-2018 National Health Interview Survey. Int J Environ Res Public Health. 2023 Apr 3;20(7):5369. doi: 10.3390/ijerph20075369. PMID 37047983
- [Result] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143